CLINICAL TRIAL: NCT01901627
Title: A Multicenter Registry to Evaluate the Clinical Outcome of Chinese Adult Patients With Active Ankylosing Spondylitis Treated With Adalimumab in the Real World Practice
Brief Title: A Multicenter Registry of Adalimumab in Chinese Adult Patients With Active Ankylosing Spondylitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IMM-12-0115
Record Dates: First submitted 2013-05-14; First posted 2013-07-17 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Spondylitis, Ankylosing
Keywords: Spondylitis, Ankylosing; adalimumab; Prospective Studies
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adalimumab: Chinese adult patients with a diagnosis of AS who meet the requirements per the local label for treatment with adalimumab.

SUMMARY:
A multicenter registry to explore the clinical outcome of Chinese adult patients with active Ankylosing Spondylitis *AS* treated with adalimumab,prescribed according to the local label,in the real world practice

DETAILED DESCRIPTION:
This registry will be conducted in a non-interventional setting for AS patients using adalimumab in China.The primary objective is to evaluate the effectiveness and safety of adalimumab in Chinese AS patients in real world clinical practice.The secondary objective is to 1)compare the clinical outcome in patients with or without good persistence with adalimumab;2)investigate the predicting factors of a good clinical response after discontinuation of adalimumab.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with established diagnosis of ankylosing spondylitis.
2. Patients eligible to use adalimumab according to the local label without any contraindication.(According to the local label, patients should be screened for active infection,TB,HBV,malignancy and CHF before the prescription of adalimumab,patients with latent TB should start a full course of anti-TB therapy before the use of adalimumab.)

Exclusion Criteria:

1.Patients with contraindication or are not appropriate to use adalimumab according to the local label will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of ankylosing spondylitis(any disease duration) who meet the requirements per the local label for treatment with adalimumab.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of adalimumab, measured as percentage of patients achieving Bath Ankylosing Spondylitis Disease Activity Index *BASDAI* 50 at week12 with adalimumab treatment. | week12

SECONDARY OUTCOMES:
Effectiveness of adalimumab measured as change in BASDAI,Ankylosing Spondylitis Disease Activity Scores *ASDAS*,Visual Analogue Scale *VAS* in pain,Patient Global Assessment *PtGA* with adalimumab treatment. | week 12
Proportion of patients who achieve each of the ASDAS disease state categories(inactive,mild,moderate,high) with adalimumab treatment. | week 12
Improvement of extra-articular manifestation with adalimumab treatment compared to baseline: uveitis flare rates, patient proportion with VAS scale at 1 in IBD PtGA, patient proportion with skin lesion clear or almost clear in psoriasis PGA. | week 12
  Physician Global Assessment*PGA*. Inflammatory Bowel Disease *IBD*
BASDAI50 response rate at week 26 and week52 in patients still on adalimumab compared to patients who discontinued adalimumab early. | week26 and 52
Change in BASDAI, ASDAS, and VAS in pain and PtGA in patients still on adalimumab compared to patients who discontinued adalimumab early. | week 26 and 52
Factors influencing the clinical response evaluated by the relapse rate(defined as BASDAI≥4) after discontinuation of adalimumab in patients who achieved BASDAI <4 and do not restart biologics in the follow-up | week 52

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China